CLINICAL TRIAL: NCT04395989
Title: An Umbrella Trial Based on Molecular Pathway for Patients With Unresectable Locally Advanced or Metastatic Triple Negative Breast Cancer (FUTURE SUPER)
Brief Title: An Umbrella Trial Based on Molecular Pathway for Patients With Metastatic TNBC.
Acronym: FUTURE-SUPER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N031
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: TNBC; Molecular Subtype; Precision Treatment; Umbrella Trial; First Line
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; famitinib; camrelizumab; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LAR-HER2mut (Experimental): If patients were LAR subtype with HER2 gene activated mutation
  Interventions: Drug: A1: Pyrotinib with nab-paclitaxel; Drug: A2: nab-paclitaxel
- LAR-PI3K/AKTmut (Experimental): If patients were LAR subtype without HER2 gene activated mutation, but had PI3K/AKT/mTOR pathway mutation
  Interventions: Drug: B1: everolimus with nab-paclitaxel; Drug: B2: nab-paclitaxel
- IM (Experimental): If patients were IM subtype (CD8 positive T cell more than 10%)
  Interventions: Drug: C1: PD-1 with nab-paclitaxel and famitinib; Drug: C2: nab-paclitaxel
- BLIS/MES-PI3K/AKTWT (Experimental): If patients were BLIS subtype or MES subtype without PI3K/AKT/mTOR pathway activation
  Interventions: Drug: D1: VEGFR and nab-paclitaxel, with maintenance of VEGFR and capecitabine; Drug: D2: nab-paclitaxel, with maintenance of capecitabine
- MES-PI3K/AKTmut (Experimental): If patients were MES subtype and had PI3K/AKT/mTOR pathway activation
  Interventions: Drug: E1: everolimus with nab-paclitaxel; Drug: E2: nab-paclitaxel

INTERVENTIONS:
Drug: A1: Pyrotinib with nab-paclitaxel — A1: pyrotinib(EGFR-TKI) 400mg po qd + nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Other Names: SHR1258
  Arms: LAR-HER2mut
Drug: A2: nab-paclitaxel — A2: nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Arms: LAR-HER2mut
Drug: B1: everolimus with nab-paclitaxel — B1: everolimus 10mg po qd + nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Arms: LAR-PI3K/AKTmut
Drug: B2: nab-paclitaxel — B2: nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Arms: LAR-PI3K/AKTmut
Drug: C1: PD-1 with nab-paclitaxel and famitinib — C1: PD-1 antibody SHR1210 200mg d1,15 ivgtt + nab-paclitaxel 100mg/m2 d1,8,15 ivgtt + famitinib 20mg po qd, 4 weeks as a cycle
  Other Names: Camrelizumab; SHR1210
  Arms: IM
Drug: C2: nab-paclitaxel — C2: nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Arms: IM
Drug: D1: VEGFR and nab-paclitaxel, with maintenance of VEGFR and capecitabine — D1: VEGFR bevacizumab 10mg/kg d1,15 ivgtt + nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle. Capecitabine with bevacizumab maintenance if intolerable toxicity was observed with no progression. Capecitabine maintenance 1000mg/m2 po bid d1-d14 every 3 weeks and bevacizumab 10mg/kg d1,15 ivgtt every 4 weeks.
  Other Names: Bevacizumab (BP102)
  Arms: BLIS/MES-PI3K/AKTWT
Drug: D2: nab-paclitaxel, with maintenance of capecitabine — D2: nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle. Capecitabine maintenance if intolerable toxicity was observed with no progression. Capecitabine maintenance 1000mg/m2 po bid d1-d14 every 3 weeks.
  Arms: BLIS/MES-PI3K/AKTWT
Drug: E1: everolimus with nab-paclitaxel — E1: everolimus 10mg po qd + nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Arms: MES-PI3K/AKTmut
Drug: E2: nab-paclitaxel — E2: nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle
  Arms: MES-PI3K/AKTmut

SUMMARY:
This is a Phase II, open-label, randomized controlled umbrella trial evaluating the efficacy and safety of multiple targeted treatment in patients with metastaticTNBC.

DETAILED DESCRIPTION:
This is a Phase II, open-label, randomized controlled umbrella trial evaluating the efficacy and safety of multiple targeted treatment vs. traditional chemotherapy in patients with unresectable locally advanced or metastatic triple negative breast cancer. The specific grouping of patients' depends on FUSCC 500+ gene panel testing and IHC subtype staining.These tests would be done on their rebiopsy tumor specimen. Specifically, as to TNBC molecular subtyping,FUSCC data identified the genomic aberrations that drive each TNBC subtype by applying an integrative analysis combining somatic mutation, copy number aberrations (CNAs) and gene expression profiles, which classified TNBC patients into four subtypes, namely luminal androgen receptor (LAR), immunomodulatory (IM), basal-like immune suppressed (BLIS), and mesenchymal-like (MES). Then, FUSCC conducted a IHC subtyping model to replace complex genomic sequencing, which have been validated in FUSCC cohort.FUSCC 500+ gene panel was developed combining public database(TCGA, METABRIC, 560WES, MSKCC-IMPACT ect.) and FUSCC private TNBC database.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1
* Expected lifetime of not less than three months
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Cancer stage: recurrent or metastatic breast cancer; Local recurrence be confirmed by the researchers could not be radical resection.
* Adequate hematologic and end-organ function, laboratory test results, obtained within 14 days prior to initiation of study treatment.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* Patients had received no previous chemotherapy or targeted therapy for metastatic triple-negative breast cancer
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm
* Have the cognitive ability to understand the protocol and be willing to participate and to be followed up.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Active or history of autoimmune disease or immune deficiency
* Active hepatitis B or hepatitis C
* Significant cardiovascular disease
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Treatment with taxel-based chemotherapy within 6 months
* Treatment with chemotherapy, radiotherapy,immunotherapy or surgery (outpatient clinic surgery excluded)within3 weeks prior to initiation of study treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Previous received anti-VEGFR small molecule tyrosine kinase inhibitors (e.g. famitinib, sorafenib, Sunitinib, regorafenib, etc.) for treatment of the patients .
* A history of bleeding, any serious bleeding events.
* Important blood vessels around tumors has been infringed and high risk of bleeding.
* Long-term unhealing wound or incomplete healing of fracture
* Urine protein ≥2+ and 24h urine protein quantitative > 1 g.
* Arrhythmia for long-term use of anti-arrhythmic drugs and New York heart association class II or higher cardiac insufficiency

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | approximately 3 years
  Refers to the time between the patient's enrollment and any recorded tumor progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | approximately 3 years
  Refers to the period from the date of the first study dose to the date of death for any reason.
Objective response rate (ORR) | approximately 3 years
  Defined as the proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time, including cases of CR and PR.
Duration of Response (DoR) | approximately 3 years
  Defined as the date from the first recording of tumor response (assessed according to RECIST 1.1) to the first recording of the objective progression of the tumor (assessed according to RECIST 1.1) or to the date of death for any reason, whichever occurs first.
Disease Control Rate (DCR) | approximately 3 years
  The proportion of subjects who received treatment and whose best overall response (BOR) was assessed as complete response (CR), partial response (PR) and stable disease (SD) ≥4 weeks according to RECIST1.1.
Safety: Adverse Events (AE) | approximately 3 years
  AE refers to any untoward medical occurrence in a study subject administered an investigational product which does not necessarily have a causal relationship with the treatment. AE is assessed according to the NCI-CTC AE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fan L, Wang ZH, Ma LX, Wu SY, Wu J, Yu KD, Sui XY, Xu Y, Liu XY, Chen L, Zhang WJ, Jin X, Xiao Q, Shui RH, Xiao Y, Wang H, Yang YS, Huang XY, Cao AY, Li JJ, Di GH, Liu GY, Yang WT, Hu X, Xia Y, Liang QN, Jiang YZ, Shao ZM. Optimising first-line subtyping-based therapy in triple-negative breast cancer (FUTURE-SUPER): a multi-cohort, randomised, phase 2 trial. Lancet Oncol. 2024 Feb;25(2):184-197. doi: 10.1016/S1470-2045(23)00579-X. Epub 2024 Jan 8. PMID 38211606